CLINICAL TRIAL: NCT03964779
Title: Prevalence of Thyroid Dysfunction and Anti-thyroid Antibodies in Infertile Women
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed M Maged, MD, professor, Cairo University
Other Study IDs: 57
Record Dates: First submitted 2019-05-23; First posted 2019-05-28 (Actual); Last update posted 2019-05-28 (Actual); Status verified 2019-05

CONDITIONS: Infertility, Female
MeSH Terms: conditions — Infertility, Female | interventions — Serum Bactericidal Antibody Assay

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Anovulatory women: 40 infertile women with either unexplained or anovulatory infertility with/without associated male factor of infertility
  Interventions: Diagnostic Test: Hormonal assay; Diagnostic Test: Antibody assay
- Tubal factor women: 40 infertile women with tubal (mechanical) factor of infertility with/without associated male factor of infertility
  Interventions: Diagnostic Test: Hormonal assay; Diagnostic Test: Antibody assay
- male factor couple: 40 women with exclusive male factor of infertility and will be used as a control group
  Interventions: Diagnostic Test: Hormonal assay; Diagnostic Test: Antibody assay

INTERVENTIONS:
Diagnostic Test: Hormonal assay — Measurement of Thyroid stimulating hormone
  Other Names: TSH assay
Diagnostic Test: Antibody assay — antithyroglobulin and antithyroid peroxidase
  Other Names: antithyroid antibodies

SUMMARY:
The study population will be divided into three groups:

* Group (A) consisting of 40 infertile women with either unexplained or anovulatory infertility with/without associated male factor of infertility,
* Group (B) consisting of 40 infertile women with tubal (mechanical) factor of infertility with/without associated male factor of infertility, and
* Group (C) consisting of 40 women with exclusive male factor of infertility and will be used as a control group.

  . All women will be subjected to:
* Informed consent
* Full history taking, including age, duration of infertility and whether primary or secondary
* General and pelvix examination
* Trans-vaginal ultrasonography
* Determination of hormonal profile (FSH, LH, Estradiol, Prolactin)
* Determination of ovulatory status
* Determination of of tubal patency
* Determination of presence of male factor
* Determination of TSH and antithyroid antibodies (antithyroglobulin and antithyroid peroxidase) blood levels

DETAILED DESCRIPTION:
The study population will be divided into three groups:

* Group (A) consisting of 40 infertile women with either unexplained or anovulatory infertility with/without associated male factor of infertility,
* Group (B) consisting of 40 infertile women with tubal (mechanical) factor of infertility with/without associated male factor of infertility, and
* Group (C) consisting of 40 women with exclusive male factor of infertility and will be used as a control group.

  . All women will be subjected to:
* Informed consent
* Full history taking, including age, duration of infertility and whether primary or secondary
* General and pelvix examination
* Trans-vaginal ultrasonography
* Determination of hormonal profile (FSH, LH, Estradiol, Prolactin)
* Determination of ovulatory status (by previous documented history of induction of ovulation OR previous ultrasonography OR previous estimation midluteal serum progesterone, etc …)
* Determination of of tubal patency (by previous hysterosalpingiography or laparoscopy)
* Determination of presence of male factor (by seminal fluid analysis)
* Determination of TSH and antithyroid antibodies (antithyroglobulin and antithyroid peroxidase) blood levels

ELIGIBILITY:
Inclusion Criteria:

* - Age: 18 - 38 years
* Infertile women whether due to functional, anatomical, male factors OR unexplained OR combined factors

Exclusion Criteria:

* - Age: below 18 and above 38 years
* Patients with autoimmune diseases (such as lupus and rheumatoid arthritis)
* Acute illness that require hospitalization
* Patients on the following medications: steroids, dopamine, iodine, amiodarone, lithium, donperidone, thyroid hormone, and phenytoin.
* Patients who work at night.

Ages: 20 Years to 40 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes
Study Population: 120 women with infertility will be divided into three groups:
  * Group (A) consisting of 40 infertile women with either unexplained or anovulatory infertility with/without associated male factor of infertility,
  * Group (B) consisting of 40 infertile women with tubal (mechanical) factor of infertility with/without associated male factor of infertility, and
  * Group (C) consisting of 40 women with exclusive male factor of infertility and will be used as a control group.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2019-05 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
prevalence of thyroid dysfunction among infertile women | through study completion, an average of 6 months
  prevalence of thyroid dysfunction (clinical or subclinical, hypothyroidism or hyperthyroidism) among infertile women

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Maged, Principal Investigator — Professor
Locations (1):
- Kasr Alainy medical school, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided